CLINICAL TRIAL: NCT03104725
Title: Does N-Acetylcysteine Decrease Spontaneous Oxidation of Central Neural Dopamine in Parkinson's Disease?
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficulty with recruitment and participant accrual due to study eligibility criteria and required study procedures (e.g., multiple lumbar punctures).
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 170076; 17-N-0076
Record Dates: First submitted 2017-04-04; First posted 2017-04-07 (Actual); Results first posted 2021-05-19 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2020-03

CONDITIONS: Parkinson Disease; Cerebrospinal Fluid
Keywords: 5-S-Cysteinyldopamine; Cerebrospinal Fluid; PARKINSONS DISEASE; MONOAMINE OXIDASE INHIBITOR
MeSH Terms: conditions — Parkinson Disease | interventions — Acetylcysteine; Spinal Puncture

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Healthy Volunteers (Experimental): HVs who undergo 2 LPs as inpatients, with 48 hours between LPs and no NAC treatment
  Interventions: Procedure: Lumbar Puncture; Radiation: Fluoroscopy
- PD Patients (Experimental): Patient undergoes a lumbar puncture (LP) as an inpatient at the NIH Clinical Center to obtain cerebrospinal fluid (CSF) for assays of Cys-DA, 3,4- dihydroxyphenylacetic acid (DOPAC), and related biochemicals. The second LP is done after the patient has taken at least 5 doses of NAC (2 grams orally twice per day).
  Interventions: Drug: N-Acetylcysteine; Procedure: Lumbar Puncture; Radiation: Fluoroscopy

INTERVENTIONS:
Drug: N-Acetylcysteine — Oral
  Arms: PD Patients
Procedure: Lumbar Puncture — Each participant undergoes a baseline lumbar puncture (LP 1) as an inpatient at the NIH Clinical Center to obtain cerebrospinal fluid (CSF) for assays of Cys-DA, 3,4-dihydroxyphenylacetic acid (DOPAC), and related biochemicals. The second LP (LP 2) is completed after the PD participant has taken at least 5 doses of NAC (2 grams orally twice per day) and approximately 2 hours after the last NAC dose. For the HV participant, LP 2 occurs approximately 48 hours after LP 1 (no NAC administered).
Radiation: Fluoroscopy — If needed for lumbar puncture

SUMMARY:
Background:

Parkinsons disease (PD) causes slow movement, stiffness, and poor balance. Many symptoms are due to the loss of brain cells that make the brain chemical dopamine. The cells may be damaged by the breakdown of dopamine by a process called oxidation. The drug N-acetylcysteine (NAC) can act as an antioxidant. Researchers want to test if NAC can decrease the oxidation of brain dopamine in people with PD.

Objective:

To look at the effect of NAC on brain chemistry in people with PD.

Eligibility:

People ages 18 and older with PD that were diagnosed within the past 5 years. They must be taking a monoamine oxidase inhibitor.

Healthy volunteer participants ages 18 and older.

Design:

Participants will be screened with:

Medical history

Physical exam

Blood and urine tests

Participants will be hospitalized for 4 to 8 days.

On day 1, participants will have blood and urine tests. For several hours, they cannot eat or drink anything but water and their medications. Late in the morning they will have a meal.

About 2 hours later they will have a spinal tap (lumbar puncture). For this, a numbing medicine is injected into the back. A needle is inserted between the bones in the back to remove a small amount of fluid. The spinal tap may use x-rays to see inside the body.

After the spinal tap, they will start taking NAC by mouth.

They will take NAC twice a day for 2 more days.

On the next day, they will not eat until a meal in the late morning. They will take a final NAC dose.

About 2 hours later they will have a second spinal tap.

Healthy Volunteer (HV) participants will receive a spinal tap on day one, followed by a second spinal tap 48 hours after the first spinal tap. HV participants will not receive NAC.

DETAILED DESCRIPTION:
Objective:

This study is to test whether N-acetylcysteine (NAC) inhibits the spontaneous oxidation of central neural dopamine as indicated by the cerebrospinal fluid (CSF) concentration of 5-S-cysteinyl-dopamine (Cys-DA) in patients with Parkinsons disease (PD).

Study population:

The study population comprises up to 35 participants with early (less than or equal to 5 years from diagnosis), mild, levodopa-untreated PD and up to 6 healthy volunteer participants. The PD participants will be on an inhibitor of monoamine oxidase (MAO) that is prescribed for their disease.

Design:

The study has a two groups employing a pretest-posttest design. Each participant undergoes a lumbar puncture (LP) as an inpatient at the NIH Clinical Center to obtain cerebrospinal fluid (CSF) for assays of Cys-DA, 3,4-dihydroxyphenylacetic acid (DOPAC), and related biochemicals. For PD participants, the second LP is done after the participant has taken at least 5 doses of NAC (2 grams orally twice per day). The LP takes place about 2 hours after the last NAC dose. For HV participants the second LP takes place approximately 48 hours after the first LP.

Outcome measures:

The main outcome measure is the CSF concentration of Cys-DA. Other outcome measures are levels of other catecholamine-related neurochemicals or of indices of oxidative stress. Depending on the results, an exploratory study may be done involving NAC at 1 gram orally twice per day.

ELIGIBILITY:
* INCLUSION CRITERIA:
* PD diagnosed within the past 5 years
* Taking a monoamine oxidase (MAO) inhibitor
* Able to provide consent
* At least18 years old

EXCLUSION CRITERIA:

* Taking levodopa in any form
* Known allergy to NAC
* Already taking an anti-oxidant dietary supplement (e.g., Olive Leaf Extract, MitoQ)
* A condition that would increase risk from a lumbar puncture (e.g., symptomatic spinal stenosis or myoclonus)
* History of a post-spinal headache that required treatment with a blood patch
* On a prescribed anti-coagulant (e.g., Coumadin, Plavix)
* Pregnant or breast-feeding
* History of alcohol or drug abuse
* Any medical condition thatcould put subjects at increased risk. Potential participants are excluded who have evidence of bone marrow, liver, or kidney failure based on abnormal screening lab results.
* On a medication that could interfere with the scientific results. An example of an exclusionary drug is the catechol-O-methyltransferase inhibitor entacapone. Tricyclic anti-depressants are another type of exclusionary drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S Goldstein, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Goldstein DS, Holmes C, Sullivan P, Jinsmaa Y, Kopin IJ, Sharabi Y. Elevated cerebrospinal fluid ratios of cysteinyl-dopamine/3,4-dihydroxyphenylacetic acid in parkinsonian synucleinopathies. Parkinsonism Relat Disord. 2016 Oct;31:79-86. doi: 10.1016/j.parkreldis.2016.07.009. Epub 2016 Jul 20. PMID 27474472
- [Background] Goldstein DS, Kopin IJ, Sharabi Y. Catecholamine autotoxicity. Implications for pharmacology and therapeutics of Parkinson disease and related disorders. Pharmacol Ther. 2014 Dec;144(3):268-82. doi: 10.1016/j.pharmthera.2014.06.006. Epub 2014 Jun 16. PMID 24945828
- [Background] Goldstein DS, Jinsmaa Y, Sullivan P, Holmes C, Kopin IJ, Sharabi Y. Comparison of Monoamine Oxidase Inhibitors in Decreasing Production of the Autotoxic Dopamine Metabolite 3,4-Dihydroxyphenylacetaldehyde in PC12 Cells. J Pharmacol Exp Ther. 2016 Feb;356(2):483-92. doi: 10.1124/jpet.115.230201. Epub 2015 Nov 16. PMID 26574516
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-N-0076.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with Parkinson's disease were recruited from the NINDS Parkinsons Clinic and the Patient Recruitment and Public Liaison Office (PRPL). Healthy participants were recruited from the PRPL.
Pre-assignment Details: All participants were screened for eligibility. Eligible participants with PD underwent a baseline LP (LP 1), followed by administration of NAC, followed by post-treatment LP (LP 2). Healthy Volunteer participants underwent a baseline LP (LP 1) and follow-up LP (LP 2) 48 hours after the baseline LP.
Groups:
- Healthy Volunteers (HVs): HV participants undergo a baseline lumbar puncture (LP 1) as an inpatient at the NIH Clinical Center to obtain cerebrospinal fluid (CSF) for assays of Cys-DA, 3,4-dihydroxyphenylacetic acid (DOPAC), and related biochemicals. The second LP (LP 2) is completed within 48 hours of LP 1. No NAC treatment is administered.
- Parkinson's Disease (PD) Patients: PD participants undergo a baseline lumbar puncture (LP 1) as an inpatient at the NIH Clinical Center to obtain cerebrospinal fluid (CSF) for assays of Cys-DA, 3,4- dihydroxyphenylacetic acid (DOPAC), and related biochemicals. The second LP (LP 2) is completed after the patient has taken at least 5 doses of N-Acetylcysteine (NAC) (2 grams orally twice per day).
Period: Overall Study
Arm/Group | Healthy Volunteers (HVs) | Parkinson's Disease (PD) Patients
Started | 2 | 4
Completed | 2 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy Volunteers: HV participants undergo a baseline lumbar puncture (LP 1) as an inpatient at the NIH Clinical Center to obtain cerebrospinal fluid (CSF) for assays of Cys-DA, 3,4-dihydroxyphenylacetic acid (DOPAC), and related biochemicals. The second LP (LP 2) is completed within 48 hours of LP 1. No NAC treatment is administered.
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteers | Parkinson's Disease (PD) Patients | Total
Number analyzed (Participants) | 2 | 4 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.5 (11.7) | 65.6 (9.7) | 59.5 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Mean Percent Change in Cerebrospinal Fluid (CSF) Concentration of 5-S-cysteinyl-dopamine (Cys-DA) Pre and Post-N-acetylcysteine (NAC) Treatment
Description: Patients with Parkinson's Disease (PD) who took N-acetylcysteine (NAC), and healthy volunteers who did not take NAC, each had two separate lumbar punctures (LP 1 and LP 2) to obtain spinal fluid. The spinal fluid samples were used to measure the amount of a brain chemical called 5-S-cysteinyl-dopamine (Cys-DA). The primary outcome measure is the mean change in CSF Cys-DA levels between pre and post-NAC treatment, which is calculated as the difference of CSF Cys-DA levels at pre-treatment (LP 1) and post-treatment (LP 2) divided by CSF Cys-DA at pre-treatment (LP 1). A greater percent decrease in Cys-DA levels in the brain would suggest that NAC may contribute to a reduction in the oxidation of brain dopamine, while a smaller percent decrease would suggest that NAC had no effect on the oxidation of brain dopamine.
Time Frame: All participants underwent a baseline LP. For PD participants, the second LP occurred approximately 2 hours after the participant had taken NAC the last NAC dose. For HV participants the second LP takes place approximately 48 hours after the first LP.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Healthy Volunteers (HVs) | Parkinson's Disease (PD) Patients
Number analyzed (Participants) | 2 | 4
percent change | 45.7 (28.1) | 20.1 (14.2)

2. Secondary Outcome: Mean Ratio of Cys-DA/DOPAC Pre and Post-treatment Lumbar Puncture With and Without N-acetylcysteine (NAC)
Description: Patients with Parkinson's Disease (PD) who took N-acetylcysteine (NAC), and healthy volunteers who did not take NAC, each had two separate lumbar punctures (LPs) to obtain spinal fluid. The spinal fluid samples were used to measure the ratio of the brain chemical called 5-S-cysteinyl-dopamine (Cys-DA) to the brain chemical called 3,4-Dihydroxyphenylacetic acid (Cys-DOPAC). Dopamine has 2 possible metabolic fates or processes of degradation. One fate is the breakdown of Dopamine by an enzyme to form DOPAC. The other fate is spontaneous oxidation to form Cys-DA. The ratio of Cys-DA to DOPAC may reflect these relative fates. If NAC reduced spontaneous oxidation to Cys-DA, then the ratio Cys-DA/DOPAC ratio would decrease between LP 1 and LP 2.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Healthy Volunteers (HVs) | Parkinson's Disease (PD) Patients
Number analyzed (Participants) | 2 | 4
ratio
  Cys-DA/DOPAC LP1 | 0.12 (0.05) | 0.16 (0.10)
  Cys-DA/DOPAC LP2 | 0.05 (0.01) | 0.13 (0.08)

3. Secondary Outcome: Mean Percent Change in Cys-DA/DOPAC Between Pre and Post-treatment Lumbar Puncture With and Without N-acetylcysteine (NAC)
Description: Patients with Parkinson's Disease (PD) who took N-acetylcysteine (NAC), and healthy volunteers who did not take NAC, each had two separate lumbar punctures (LPs) to obtain spinal fluid. The spinal fluid samples were used to measure the ratio of the brain chemical called 5-S-cysteinyl-dopamine (Cys-DA) to the brain chemical called 3,4-Dihydroxyphenylacetic acid (Cys-DOPAC). Dopamine has 2 metabolic fates. One is the breakdown of dopamine by an enzyme to form DOPAC. The other is spontaneous oxidation to form Cys-DA. The ratio of Cys-DA/DOPAC may reflect these relative fates. If NAC reduced spontaneous oxidation to Cys-DA, then the ratio Cys-DA/DOPAC would decrease between LP 1 and LP 2, which would be reflected as a percent decrease.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Healthy Volunteers (HVs) | Parkinson's Disease (PD) Patients
Number analyzed (Participants) | 2 | 4
percent change | 50.1 (16.2) | 27.2 (5.0)

ADVERSE EVENTS:
Time Frame: Duration of participation in study and up to 8 days following the second LP
Arm/Group | Healthy Volunteers (HVs) | Parkinson's Disease (PD) Patients
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4
Other Adverse Events (participants affected / at risk) | 2/2 | 1/4
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Volunteers (HVs) (N=2) | Parkinson's Disease (PD) Patients (N=4)
Puncture site pain (General disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-11): https://cdn.clinicaltrials.gov/large-docs/25/NCT03104725/Prot_SAP_000.pdf